CLINICAL TRIAL: NCT00686764
Title: Evaluation of Ultrasonic Neuroma Size With Residual Limb Pain in Above Knee Amputees
Brief Title: Evaluation of Ultrasonic Neuroma Size With Residual Limb Pain in Above-Knee Amputees
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Hans Carlson, Associate professor of physical medicine and rehabilitation in the Department of Orthopaedics and Rehabilitation, Oregon Health and Science University
Other Study IDs: OHSUIRB#3862
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Neuroma Amputation
Keywords: trans-femoral amputation
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Trans-femoral amputees that meet the eligibility criteria.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Using ultrasound, we will measure the cross-sectional area of the neuroma at its widest point and compare to the cross-sectional area of the same nerve at the lesser trochanter.
  We will be using four different metrics for quantifying the pain experience of each subject: Questionnaire for Persons with Transfemoral Amputation (Q-FTA), Trinity Amputation and Prosthesis Experience Scales (TAPES), Visual Analog Scale (VAS), and the Short-Form 36 (SF-36).

SUMMARY:
Background: The formation of neuromas, a fusiform swelling of a nerve or nerve ending, is a well documented response to limb amputation. Likewise, Residual Limb Pain (RLP), pain felt from the remaining portion of the amputated limb, is common among amputees. Neuromas are found in more than 90% of lower extremity amputations, of which 30-50% are pain-generating for the patient . And while surgical techniques reveal the commonly held belief that neuroma formation is one of the causal drivers behind RLP, there has been no study to demonstrate that the two events - namely the magnitude of neuroma formation and the magnitude of pain experienced by amputees - are correlated. If this correlation, or lack thereof, were elucidated with the use of ultrasonography, this would provide the preliminary data which could lead to further studies in neuroma minimization and/or proliferation.

Objective: This study seeks to use ultrasonography (US) to quantify the degree to which neuroma size and the nature of surrounding tissue correlate with the experience of RLP in trans-femoral amputees.

Setting and Subjects: This study will enroll 30 trans-femoral amputees, male and female, who are over the age of 18. The study will take place in the OHSU Orthopaedic Outpatient Clinic, and OHSU Imaging Department.

Intervention: None. This is an observational clinical study in which we will characterize the sciatic nerve/neuroma and surrounding tissue using ultrasound.

Measurements: We will use US to measure the cross sectional area of the neuroma at its widest point and compare this to the cross section of the same neuron at the lesser trochanter. Furthermore, we will describe the morphology of the neuroma. To quantify the subject's pain experience we will utilize the Questionnaire for Persons with Transfemoral Amputation (Q-TFA), Trinity Amputation & Prosthetic Experience Scale (TAPES), Visual Analog Scale (VAS), and the Short Form 36 (SF-36).

Analysis: The statistical analysis will employ a Pearson correlation coefficient and linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years old
* a trans-femoral amputee
* more than one year post-amputation
* has worn a prosthesis within the last year

Exclusion Criteria:

* subject also diagnosed with diabetes
* subject also diagnosed with Peripheral Vascular Disease
* subject also diagnosed with peripheral neuropathy
* subject with spinal cord, head, or nerve root injury

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will consist of 25 trans-femoral amputees meeting the inclusion and exclusion criteria. We will recruit participants from the OHSU clinics, Primary Care Clinics, and specialty clinics including orthopaedic surgery, general surgery, pain centers, neurology, and orthotics and prosthesis clinics and offices. We anticipate that the majority of subjects will be recruited from the Department of Orthopaedics and Rehabilitation's clinical practice. Potential subjects will be identified from the investigators' clinic and medical records. Recruiting outside of the Department of Orthopaedics and Rehabilitation will be done using recruiting posters and letters addressed to the primary care physicians, specialists and at prosthetic clinics. Recruitment notices will be posted on the OHSU and Department of Orthopaedics and Rehabilitation's Web sites and the OHSU Study Participation Web site. We intend to enroll 30 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Ultrasonic neuroma size | Single observation at time of consent
Residual limb pain | Single observation at time of consent

CONTACTS AND LOCATIONS:
Overall Officials: Hans Carlson, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Center for Health & Healing, Portland, Oregon, United States